CLINICAL TRIAL: NCT03333369
Title: L-Dopa Modulated Striatal Functional Connectivity in Schizotypal Adults: a Randomized Double-blind Placebo-controlled Study
Brief Title: Exceptional Experiences (EE), Salience & Dopaminergic Neurotransmission
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DA_EE_Salience
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy; Schizotypal Personality
Keywords: resting-state functional MRI; Dopamine; functional connectivity
MeSH Terms: conditions — Schizotypal Personality Disorder | interventions — benserazide, levodopa drug combination; Glucose

STUDY DESIGN:
Intervention Model Description: Each subject in the group will participate in two test sessions, separated by at least one week. All sessions will start at 15:30.
  In a double-blind within-design procedure, participants will be randomly assigned to receive either a cachet of a dual-release formulation of 200 mg levodopa/50 mg benserazide (a peripheral L-dihhydroxyphenylalanine-decarboxylase inhibitor) or a placebo in the first session. In the second session they will receive the other intervention.
Who Masked: Participant, Care Provider, Investigator
Masking Description: For the randomization of the intervention and placebo the "Research Randomizer" on www.randomizer.org will be used. The randomization will be performed by the Kantonsapotheke in Zurich. The generated list of condition sequences will be stored at there. The list will not be accessible for study members who are associated with the assessment. The Boxes containing the cachets will be labelled with the subject number and A or B for the first or second session, respectively as well as with the ID of the study. The cachets will be prepared and labelled at the Kantonsapotheke in Zurich. DA and placebo will be provided in identical cachets. The blinding will be broken only after a subject has completed both experimental sessions or in case of an acute reaction during the session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Madopar Arm (Active Comparator): A single dose of a cachet filled with 200 mg levodopa/50 mg benserazide
  Interventions: Drug: 200 mg levodopa/50 mg benserazide
- Placebo Arm (Placebo Comparator): A single dose of a cachet filled with Dextrose
  Interventions: Drug: Dextrose

INTERVENTIONS:
Drug: 200 mg levodopa/50 mg benserazide
  Other Names: Madopar DR
  Arms: Madopar Arm
Drug: Dextrose
  Other Names: Placebo
  Arms: Placebo Arm

SUMMARY:
The dopamine hypothesis of schizophrenia implies that alterations in the dopamine system cause functional abnormalities in the brain that may converge to aberrant salience attribution and eventually lead to psychosis. Indeed, widespread brain disconnectivity across the psychotic spectrum has been revealed by resting-state functional magnetic resonance imaging (rs-fMRI). However, the dopaminergic involvement in intrinsic functional connectivity (iFC) and its putative relationship to the development of psychotic spectrum disorders remains partly unclear - in particular at the low-end of the psychosis continuum. Therefore, the investigators examined dopamine-induced changes in striatal iFC and their modulation by psychometrically assessed schizotypy. The randomized, double-blind placebo-controlled study design included 54 healthy, right-handed male participants. Each participant was assessed with the Schizotypal Personality Questionnaire (SPQ) and underwent 10 min of rs-fMRI scanning. Participants then received either a placebo or 200 mg of L-DOPA, a dopamine precursor. The investigators analyzed iFC of six striatal seeds that are known to evoke modulation of dopamine-related networks.

The investigators hypothesized that, within the L-DOPA treatment group, the striatal iFC would be disrupted due to increased availability of dopamine. The investigators further hypothesized that individuals with high schizotypal scores would show a disruption of striatal connectivity, as has been reported with schizophrenia. In addition, the investigators hypothesized that the L-DOPA-dependent change in striatal iFC would interact with the severity of positive symptoms, as has been found in previous studies in non-clinical psychosis. The investigators anticipated this symptom-dependent change, especially in the ventral striatal regions, because these are thought to modulate cortico-striatal loops associated with cognition and emotion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* Between 20 and 40 years of age,
* With exceptional experiences or skeptics,
* Caucasian origin,
* Normal visual and acoustic accuracy.

Exclusion Criteria:

* Persons with a personal or first-degree family history of neurological and psychiatric disease, including impaired cognitive abilities,
* Pregnant or breastfeeding women,
* Chronic or acute pain,
* Acute or chronic somatic disease,
* Women (i.e. only men included),
* Men over 40 years of age or below 20,
* left- or mixed-handedness,
* General MRI exclusion criteria,
* General Dopamine-Challenge exclusion criteria,
* Hormonal or herbal therapy,
* Smoker.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2015-08-13 (Actual); Study Completion 2015-08-13 (Actual)

PRIMARY OUTCOMES:
intrinsic functional connectivity | 2 hours
  Dopamine dependent intrinsic functional connectivity as measured by resting-state functional magnetic resonance imaging

SECONDARY OUTCOMES:
Schizotypy | 15 min
  Schizotypy scores assessed by the Schizotypal Personality Questionnaire (SPQ):
  * n of items 74 (min. score = 0 ; max. score = 74): higher score implies higher level of schizotypy
  * Subscales:
    * Cognitive Perceptual (min. score = 0 ; max. score = 33)
    * Interpersonal (min. score = 0 ; max. score = 25)
    * Disorganized (min. score = 0 ; max. score = 16)

CONTACTS AND LOCATIONS:
Locations (1):
- Collegium Helveticum, ETH & Universität Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No